CLINICAL TRIAL: NCT02736409
Title: A Phase 3, Multicenter, Double-blind Extension Study to Evaluate Maintenance of Efficacy of Oral Budesonide Suspension (OBS) and Long-term Treatment Effect of OBS in Adolescent and Adult Subjects (11 to 55 Years of Age, Inclusive) With Eosinophilic Esophagitis (EoE)
Brief Title: An Extension Study to Evaluate Maintenance of Efficacy and Long-term Treatment Effect of Oral Budesonide Suspension (OBS) in Adults and Adolescents With Eosinophilic Esophagitis (EoE)
Acronym: ORBIT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP621-302
Record Dates: First submitted 2016-03-22; First posted 2016-04-13 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2020-12

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arms A OBS Completers/ Responders (Experimental): Arm A Oral Budesonide Suspension Completers/ Responders
  Interventions: Drug: Oral Budesonide Suspension (OBS)
- Arm B OBS Completers/ Responders (Placebo Comparator): Arm B Oral Budesonide Suspension Completers/ Responders. 1:1 randomization for Arms A and B
  Interventions: Drug: Placebo
- Arm C OBS Completers/ Non-Responders (Experimental): Arm C Oral Budesonide Suspension Completers/ Non-Responders
  Interventions: Drug: Oral Budesonide Suspension (OBS)
- Arm D Placebo Completers (Experimental): Arm D Placebo Completers
  Interventions: Drug: Oral Budesonide Suspension (OBS)

INTERVENTIONS:
Drug: Oral Budesonide Suspension (OBS) — OBS 2mg twice daily
  Arms: Arm C OBS Completers/ Non-Responders; Arm D Placebo Completers; Arms A OBS Completers/ Responders
Drug: Placebo — Matching Placebo dose
  Arms: Arm B OBS Completers/ Responders

SUMMARY:
This is a multicenter, double- blind extension study of Oral Budesonide Suspension (OBS) in adults and adolescents (11 to 55 years of age, inclusive) with Eosinophilic Esophagitis (EoE) who have completed participation in the SHP621-301 induction study (NCT02605837). The primary objective is to evaluate the maintenance of efficacy of OBS over 36 weeks. Maintenance of efficacy will be measured by the peak eosinophilic count and Dysphagia Symptom Questionnaire (DSQ) score.

ELIGIBILITY:
Inclusion Criteria:

1. Subject completed SHP621-301 induction study.
2. Subject is able to provide written informed consent (subject, parent or legal guardian and, as appropriate, subject assent) to participate in the study before completing any study-related procedures.
3. Subject is male or female aged 11-55 years, inclusive, at time of consent for SHP621-301 study.
4. Subject is willing and able to continue any dietary therapy, environmental therapy, and/or medical regimens (including gastric acid suppression; see exclusions below) in effect at the screening visit (Visit 0). There should be no changes to these regimens during study participation.
5. All female subjects must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-hCG]) prior to enrollment into the study. Females of childbearing potential must agree to continue acceptable birth control measures (eg, abstinence, stable oral contraceptives, or double-barrier methods) throughout study participation and for 30 days following the last dose of investigational product.
6. Subject is willing and has an understanding and ability to fully comply with study procedures including DSQ compliance (completed the DSQ on ≥70% of days in any 2 consecutive weeks of the screening period)and restrictions defined in this protocol

Exclusion Criteria:

1. Subject has changes in medications that could affect the study or diet in the weeks since the final treatment evaluation visit (Visit 4) of the SHP621-301 study.
2. Subject using immunomodulatory therapy since the final treatment evaluation visit (Visit 4) of the SHP621-301 study or anticipated use of immunomodulatory therapy during the treatment period (except for any ongoing regimen of allergy shots); any temporary use (≤7 days) or initiation of new steroid treatment during the study should be documented and discussed with the medical monitor prospectively but cannot occur within 4 weeks of scheduled EGDs.
3. Subject using swallowed topical corticosteroid for EoE or systemic corticosteroid for any condition since the final treatment evaluation visit (Visit 4) of the SHP621-301 study or anticipated use during the treatment period; any temporary use (≤7 days) or initiation of new steroid treatment during the study should be documented and discussed with medical monitor prospectively but cannot occur within the 4 weeks of the scheduled EGDs.
4. Subject on inhaled or intranasal steroids and not on a stable dose between the baseline visit (Visit 1) of the SHP621-301 study and the screening EGD of this study.
5. Subject has initiated, discontinued, or changed dosage regimen of proton pump inhibitors (PPIs), H2 antagonists, antacids, antihistamines, or leukotriene inhibitors for any condition (such as gastroesophageal reflux disease, asthma or allergic rhinitis) since the final treatment evaluation visit (Visit 4) of the SHP621-301 study or anticipated changes in the use of such medications during the treatment period.
6. Subject using Cytochrome P450 3A4 inhibitors (eg, ketoconazole, grapefruit juice) since the final treatment evaluation visit (Visit 4) of the SHP621-301 study or anticipated use of such medications during the treatment period.
7. Subject has an appearance on screening EGD of an esophageal stricture (high grade), as defined by the presence of a lesion that does not allow passage of a diagnostic adult upper endoscope (eg, with an insertion tube diameter of >9mm).
8. Subject is on a pure liquid diet or the six-food elimination diet.
9. Subject has presence of esophageal varices at the EGD at the final treatment evaluation visit (Visit 4) of the SHP621-301 study.
10. Subject has any current disease of the gastrointestinal tract, aside from EoE, including eosinophilic gastritis, enteritis, colitis, or proctitis, inflammatory bowel disease, or celiac disease.
11. Subject has other diseases causing or associated with esophageal eosinophilia, including hypereosinophilic syndrome, collagen vascular disease, vasculitis, achalasia, or parasitic infection.
12. Subject has oropharyngeal or esophageal candidiasis that failed to respond to previous treatment.

    Diagnosis with oropharyngeal or esophageal candidiasis at or since the final treatment evaluation visit (Visit 4) of the SHP621-301 study is not an exclusion as long as the subject received treatment for candidiasis and is expected to respond to treatment.
13. Subject has acute or chronic infection or immunodeficiency condition, including tuberculosis, fungal, bacterial, viral/parasite infection, ocular herpes simplex, or chicken pox/measles.
14. Subject has upper gastrointestinal bleeding identified in the EGD at the final treatment evaluation visit (Visit 4) of the SHP621-301 study or since the final treatment evaluation visit (Visit 4) of the SHP621-301 study.
15. Subject has evidence of active infection with Helicobacter pylori.
16. Subject has evidence of unstable asthma since the final treatment evaluation visit (Visit 4) of the SHP621-301 study.
17. Subject is female and pregnant or nursing.
18. Subject has a history of intolerance, hypersensitivity, or idiosyncratic reaction to budesonide (or any other corticosteroids), or to any other ingredients of the study medication.
19. Subject has a history or high risk of noncompliance with treatment or regular clinic visits.
20. Subject is on sucralfate or anticipates using sucralfate during the treatment period.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (62):
- United States (62):
  - Children's Hospital, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology, Lone Tree, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Connecticut GI, PC - Research Division, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nature Coast Clinical Research LLC, Inverness, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois College of Medicine at Peoria Pediatric Subspecialty Clinic, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Aquiant Research, New Albany, Indiana
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Clinical Trials of America LA LLC - PPDS, West Monroe, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Minnesota Gastroenterology PA, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Mount Sinai Medical Center, New York, New York
  - Asheville Gastroenterology Associates PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Clinical Trials of America-NC, LLC - PPDS, Mount Airy, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Gastrointestinal and Liver Diseases Consultants PC, Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- [Derived] Dellon ES, Collins MH, Katzka DA, Mukkada VA, Falk GW, Zhang W, Goodwin B, Terreri B, Boules M, Desai NK, Hirano I. Effect of randomized treatment withdrawal of budesonide oral suspension on clinically relevant efficacy outcomes in patients with eosinophilic esophagitis: a post hoc analysis. Therap Adv Gastroenterol. 2024 Dec 23;17:17562848241307602. doi: 10.1177/17562848241307602. eCollection 2024. PMID 39735351
- [Derived] Dellon ES, Collins MH, Katzka DA, Mukkada VA, Falk GW, Morey R, Goodwin B, Eisner JD, Lan L, Desai NK, Williams J, Hirano I; ORBIT2/SHP621-302 Investigators. Long-Term Treatment of Eosinophilic Esophagitis With Budesonide Oral Suspension. Clin Gastroenterol Hepatol. 2022 Jul;20(7):1488-1498.e11. doi: 10.1016/j.cgh.2021.06.020. Epub 2021 Jun 26. PMID 34182150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 70 sites in United States from 01 April 2016 (first participant enrolled) to 12 November 2019 (last participant completed).
Pre-assignment Details: A total of 219 participants who completed the study SHP621-301 (NCT02605837) and consented to participate in the current study SHP621-302 (NCT02736409) were enrolled and received at least one dose of investigational product (IP), among which 174 participants completed this study .
Groups:
- Full Responder BOS-PBO Group: Full responder BOS (Budesonide Oral Suspension)-PBO (Placebo) group consisted of participants who were full responders at the end of 12 weeks double-blind treatment with BOS in SHP621-301 (NCT02605837) and who were randomized to double-blind placebo twice daily. Participants received 10 milliliter (mL) of 0.2 milligram per milliliter (mg/mL) placebo orally twice daily for 36 weeks.
- Full Responder BOS-BOS Group: Full responder BOS-BOS group consisted of participants who were full responders at the end of 12 weeks double-blind treatment with BOS in SHP621-301 (NCT02605837) and who were randomized to remain on double-blind BOS 2 mg twice daily. Participants received 10 mL of 0.2 mg/mL BOS twice daily for 36 weeks.
- Non-Responder BOS-BOS Group: Non-responder BOS-BOS group consisted of participants who were not full responders (ie, partial or non-responders) at the end of 12 weeks double-blind treatment with BOS in SHP621-301 (NCT02605837) and who continued to receive double-blind BOS 2 mg twice daily. Participants received 10 mL of 0.2 mg/mL BOS twice daily for 36 weeks.
- PBO-BOS Group: PBO-BOS group consisted of participants who received placebo in SHP621-301 (NCT02605837) and were assigned to receive double-blind BOS 2 mg twice daily. Participants received 10 mL of 0.2 mg/mL BOS twice daily for 36 weeks.
Period: Overall Study
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Started | 23 | 25 | 106 | 65
Completed | 19 | 22 | 80 | 53
Not Completed | 4 | 3 | 26 | 12
Not completed — Withdrawal by Subject | 4 | 2 | 17 | 3
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 5 | 4
Not completed — Other | 0 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all randomized participants who received at least 1 dose of investigational product in the NCT02736409 (SHP621-302) study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group | Total
Number analyzed (Participants) | 23 | 25 | 106 | 65 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (11.66) | 36.8 (14.09) | 33.1 (12.02) | 33.5 (12.61) | 34.0 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 42 | 26 | 86
  Male | 16 | 14 | 64 | 39 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 1 | 5
  Not Hispanic or Latino | 23 | 25 | 101 | 62 | 211
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 4 | 0 | 5
  White | 22 | 24 | 95 | 62 | 203
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 6 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Had Relapse During the Entire Week 36 Period
Description: Relapse (Yes/No) was defined as meeting both the eosinophil histology relapse criterion and the dysphagia symptom relapse criterion. Eosinophil histology relapse was defined as an eosinophil count of greater than or equal to(> or =) 15 per high-power field (eos/hpf) from at least 2 of 3 levels of the esophagus. Dysphagia symptom relapse was defined as having at least 4 days of dysphagia (with answer 'Yes' for question 2 in DSQ [Dysphagia Symptom Questionnaire]) in the 2-week period prior to the scheduled visit, as determined by the DSQ.
Time Frame: Week 36
Population: SHP621-301 (NCT02605837) BOS Full Responder FAS consisted of all randomized participants who were determined to be Full responders to the BOS treatment during the induction study SHP621-301 (NCT02605837) and who received at least 1 dose of IP in the SHP621-302 (NCT02736409) study.
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group
Number analyzed (Participants) | 23 | 25
proportion of participants | 0.43 | 0.24
Statistical Analysis 1: Comparison: Full Responder BOS-PBO Group vs Full Responder BOS-BOS Group; Test type: Superiority; p = 0.131, Fisher Exact; Difference in Proportion = -0.19, 95% CI 2-sided [-0.452 to 0.082]

2. Secondary Outcome: Proportion of Participants With Long-term Treatment Response From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: Long-term response from SHP621-301 baseline defined: histologic response,defined as peak eosinophil count of less than or equal to(< or =)6/HPF across all available esophageal levels at Week 36 and Dysphagia symptom response 1,defined as >or= 30 percent(%) reduction in DSQ combined score(Questions [Q] 2+3) from baseline of SHP621-301 to Week 36.DSQcontain 4 questions,all participants used diary,responded to Q1(didyoueatsolid food),Q2(did food pass slowly or get stuck). If participant's answer to Q2 was No,diary ended for day. If participant answered Yes,he/she advanced to Q3(didyouhavetodoanything to make food go downorget relief), Q4(extent to which participant experienced pain while swallowing).DSQ combined score= ([sum of points from Q2+3 in daily DSQ]×14)/Number of diaries reported with non-missing data.Scale range was0-2 forQ2 and 0-4 forQ 3.Scale range for DSQ combined score was 0-84.Highervaluesrepresentingworseoutcome.Negative change from baseline indicates symptoms decreased.
Time Frame: Week 36
Population: SHP621-301 (NCT02605837) BOS Non responder FAS included all randomized participants who did not respond or partially responded to assigned BOS treatment in the induction study SHP621-301 (NCT02605837) and who received at least 1 dose of IP in the SHP621-302 (NCT02736409) study.
Measure: Number; unit: proportion of participants
Arm/Group | Non-Responder BOS-BOS Group
Number analyzed (Participants) | 106
proportion of participants | 0.13

3. Secondary Outcome: Proportion of Participants With Long-term Treatment Response From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: Long-term response from baseline defined: histologic response, defined as peak eosinophil count of less than or equal to(< or =) 6/HPF across all available esophageal levels at Week 36 and Dysphagia symptom response 1,defined as >or= 30 percent(%) reduction in DSQ combined score (Questions [Q] 2+3) from baseline of SHP621-301 to Week 36.DSQcontain 4 questions,all participants used diary,responded to Q1(did you eat solid food),Q2(did food pass slowly or get stuck). If participant's answer to Q2 was No,diary ended for day. If participant answered Yes,he/she advanced to Q3(didyouhavetodoanything to make food go downorget relief), Q4(extent to which participant experienced pain while swallowing).DSQ combined score= ([sum of points from Q2+3 in daily DSQ]×14)/Number of diaries reported with non-missing data.Scale range was0-2 forQ2 and 0-4 forQ 3.Scale range for DSQ combined score was 0-84. Higher values representing worse outcome.Negative change from baseline indicates symptoms decreased.
Time Frame: Week 36
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Non-Responder BOS-BOS Group
Number analyzed (Participants) | 106
proportion of participants | 0.06

4. Secondary Outcome: Proportion of Participants Who Had a Histologic Response (Eosinophil Count of Less Than or Equal to (<or=6)/High-Powered Field [HPF]) at Week 12 and Week 36
Description: Histology response was defined as a peak eosinophil count of <or=6/HPF across all available levels at Week 12 and Week 36.
Time Frame: Week 12 and Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study.
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.04 | 0.76 | 0.27 | 0.57
  Week 36 | 0.30 | 0.52 | 0.21 | 0.38

5. Secondary Outcome: Proportion of Participants Who Had at Least a 30 Percent (%) Change in DSQ Combined Score From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 12 and Week 36
Description: Dysphagia symptom response with respect to the baseline of induction study (SHP621-301 [NCT02605837]) was defined as 30% reduction in DSQ combined score (questions 2+3) at Week 12 and Week 36 of current study from baseline of the induction study. DSQ contain 4 questions, all participants used a diary and responded to Q1 (did you eat solid food), Q2 (did food pass slowly or get stuck). If participant's answer to Q2 was No, then diary ended for that day. If participant answered Yes,he/she advanced to Q3 (did you have to do anything to make food go down or get relief) and Q4 (extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ] × 14)/Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q3. Scale range for DSQ combined score was 0-84. Higher values representing worse outcome. Negative change from baseline indicates symptoms decreased.
Time Frame: Baseline of SHP621-301 (NCT02605837), Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.74 | 0.84 | 0.47 | 0.57
  Week 36 | 0.78 | 0.84 | 0.46 | 0.58

6. Secondary Outcome: Proportion of Participants Who Had at Least a 30 Percent (%) Change in DSQ Combined Score From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 12 and Week 36
Description: Dysphagia symptom response with respect to the baseline of current study (SHP621-302 [NCT02736409]) was defined as 30% reduction in DSQ combined score (questions 2+3) at Week 12 and Week 36 from baseline of the current study. DSQ contain 4 questions, all participants used diary and responded to Q1 (did you eat solid food), Q2 (did food pass slowly or get stuck). If participant's answer to Q2 was "No", then diary ended for that day. If participant answered "Yes",he/she advanced to Q3 (did you have to do anything to make food go down or get relief) and Q4 (extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ] × 14)/Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q 3. Scale range for DSQ combined score was 0-84. Higher values representing a worse outcome. A Negative change from baseline indicates symptoms decreased.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.13 | 0.44 | 0.24 | 0.43
  Week 36 | 0.39 | 0.40 | 0.25 | 0.42

7. Secondary Outcome: Change From Induction Study (SHP621-301 [NCT02605837]) Baseline in Total Endoscopy Score at Week 12 and Week 36 of Current Study
Description: Endoscopic findings with separate evaluations of the proximal and distal esophagus were recorded with respect to 5 categories: 1) exudates or plaques (grade 0-2); 2) fixed esophageal rings (grade 0-3); 3) edema (grade 0-2); 4) furrows (grade 0-2); and 5) strictures (grade 0-1). An endoscopy score for each category was calculated and summed for each anatomic location (proximal and distal). The minimum and maximum endoscopy score was 0 and 10 points respectively for each location (proximal and distal) and the total endoscopy score was the sum of the scores for the proximal and distal locations (maximum total score of 20 points respectively). The higher score indicated worse appearance. A negative change from baseline indicates that appearance improved.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 12 and Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study. Here the number of participants analyzed signifies participants who had an evaluable Induction Study (SHP621-301 [NCT02605837]) baseline and assessment at specific category/time point.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
Score on scale
  Week 12: number analyzed (Participants) | 20 | 24 | 91 | 59
  Week 12 | -1.9 (0.51) | -5.3 (0.69) | -3.8 (0.43) | -4.7 (0.46)
  Week 36: number analyzed (Participants) | 19 | 22 | 79 | 52
  Week 36 | -2.7 (0.60) | -4.2 (0.84) | -4.3 (0.47) | -4.4 (0.46)

8. Secondary Outcome: Change From Current Study (SHP621-302 [NCT02736409]) Baseline in Total Endoscopy Score at Week 12 and Week 36
Description: as for outcome 7
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 12 and Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study. Here the number of participants analyzed signifies participants who had an evaluable current Study (SHP621-302 [NCT02736409]) baseline and assessment at specific category/time point.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
Score on scale
  Week 12: number analyzed (Participants) | 20 | 24 | 91 | 59
  Week 12 | 0.7 (0.67) | -1.0 (0.69) | -0.3 (0.28) | -2.6 (0.46)
  Week 36: number analyzed (Participants) | 19 | 22 | 79 | 52
  Week 36 | 0.2 (0.70) | 0.0 (0.70) | -0.6 (0.34) | -2.3 (0.57)

9. Secondary Outcome: Change From Induction Study (SHP621-301 [NCT02605837]) Baseline in Peak Eosinophil Count at Week 12 and Week 36 of Current Study
Description: Change from induction study (SHP621-301 [NCT02605837]) baseline in peak eosinophil count at Week 12 and Week 36 of current study was reported.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 12 and Week 36
Population: as for outcome 7
Measure: Mean (Standard Error); unit: eosinophil count
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
eosinophil count
  Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Week 12 | -20.8 (13.41) | -60.1 (9.26) | -33.2 (5.14) | -70.3 (7.74)
  Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Week 36 | -59.8 (13.24) | -40.3 (13.23) | -33.2 (5.50) | -57.2 (7.68)

10. Secondary Outcome: Change From Current Study (SHP621-302 [NCT02736409]) Baseline in Peak Eosinophil Count at Week 12 and Week 36
Description: Change from current study (SHP621-302 [NCT02736409]) baseline in peak eosinophil count at Week 12 and Week 36 was reported.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 12 and Week 36
Population: as for outcome 8
Measure: Mean (Standard Error); unit: eosinophil count
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
eosinophil count
  Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Week 12 | 66.0 (11.52) | 7.5 (3.56) | 7.6 (3.95) | -54.4 (5.65)
  Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Week 36 | 25.5 (7.83) | 26.9 (11.18) | 6.8 (4.63) | -39.1 (6.94)

11. Secondary Outcome: Proportion of Participants Who Had Peak Eosinophil Count Less Than (<) 15/High-Powered Field (HPF) at Week 12 and Week 36
Description: Proportion of participants who had Peak Eosinophil Count less than (<) 15/HPF at Week 12 and Week 36 were reported.
Time Frame: Week 12 and Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure at specific category.
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.13 | 0.76 | 0.37 | 0.63
  Week 36 | 0.52 | 0.60 | 0.29 | 0.42

12. Secondary Outcome: Proportion of Participants Who Had Peak Eosinophil Count Less Than or Equal to (< or =) 1/High-Powered Field (HPF) at Week 12 and Week 36
Description: Proportion of participants who had Peak Eosinophil Count less than or equal to (< or =) 1/High-Powered Field (HPF) at Week 12 and Week 36 were reported.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.00 | 0.60 | 0.15 | 0.42
  Week 36 | 0.13 | 0.44 | 0.14 | 0.26

13. Secondary Outcome: Change From Induction Study (SHP621-301 [NCT02605837]) Baseline in Peak Eosinophil Count for Each Available Esophageal Level (Proximal, Mid, and Distal) at Week 12 and Week 36 of Current Study
Description: Change from induction study (SHP621-301 [NCT02605837]) baseline in peak eosinophil count for each available esophageal level (proximal, mid, distal) at Week 12 and Week 36 of current study were reported.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 12 and Week 36
Population: FAS included all randomized participants who received at least one dose of a SHP621-302 (NCT02736409) investigational product. Here the number of participants analyzed signifies participants who had an evaluable Induction Study (SHP621-301 [NCT02605837]) baseline and assessment at specific category/time point.
Measure: Mean (Standard Error); unit: eosinophil count
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
eosinophil count
  Proximal: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Proximal: Week 12 | -9.2 (13.96) | -23.3 (4.94) | -24.0 (4.38) | -41.6 (6.65)
  Proximal: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Proximal: Week 36 | -21.0 (7.09) | -19.6 (6.43) | -24.2 (4.44) | -42.3 (7.03)
  Mid: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Mid: Week 12 | -14.8 (10.80) | -53.4 (9.85) | -32.7 (4.80) | -53.8 (6.16)
  Mid: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Mid: Week 36 | -36.8 (9.89) | -47.7 (9.21) | -29.1 (5.05) | -40.8 (7.01)
  Distal: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 56
  Distal: Week 12 | -17.1 (12.11) | -44.0 (6.74) | -23.0 (5.17) | -53.6 (6.64)
  Distal: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 51
  Distal: Week 36 | -51.2 (13.69) | -25.3 (12.45) | -26.4 (5.38) | -40.2 (7.71)

14. Secondary Outcome: Change From Current Study (SHP621-302 [NCT02736409]) Baseline in Peak Eosinophil Count for Each Available Esophageal Level (Proximal, Mid, and Distal) at Week 12 and Week 36
Description: Change from current study (SHP621-302 [NCT02736409]) baseline in peak eosinophil count for each available esophageal level (proximal, mid, distal) at Week 12 and Week 36 were reported.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 12 and Week 36
Population: FAS included all randomized participants who received at least one dose of a SHP621-302 (NCT02736409) investigational product. Here the number of participants analyzed signifies participants who had an evaluable current Study (SHP621-302 [NCT02736409]) baseline and assessment at specific category/time point.
Measure: Mean (Standard Error); unit: eosinophil count
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
eosinophil count
  Proximal: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Proximal: Week 12 | 26.5 (10.44) | 2.8 (2.14) | 6.5 (2.92) | -30.8 (4.73)
  Proximal: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Proximal: Week 36 | 10.0 (3.95) | 6.9 (4.68) | 6.8 (3.25) | -23.1 (4.91)
  Mid: Week 12: number analyzed (Participants) | 19 | 24 | 90 | 57
  Mid: Week 12 | 38.4 (10.50) | 5.4 (2.88) | 3.2 (4.20) | -41.4 (5.55)
  Mid: Week 36: number analyzed (Participants) | 18 | 22 | 79 | 52
  Mid: Week 36 | 17.9 (7.72) | 12.5 (6.81) | 7.3 (4.50) | -28.9 (7.00)
  Distal: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Distal: Week 12 | 55.8 (10.04) | 7.3 (3.51) | 7.8 (3.66) | -41.6 (5.09)
  Distal: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Distal: Week 36 | 21.3 (6.47) | 24.2 (10.50) | 4.4 (4.03) | -29.5 (6.20)

15. Secondary Outcome: Change From Induction Study (SHP621-301 [NCT02605837]) Baseline in the Histopathologic Epithelial Features Combined Total Score (Grade and Stage) at Week 12 an Week 36 of Current Study
Description: Eight histopathologic epithelial features (basal layer hyperplasia, eosinophil peak, abscesses, surface layering, dilated intercellular spaces, surface alteration, dyskeratotic epithelial cells, lamina propria fibrosis) are scored on a 4-point scale (0=normal, 3=worst) for both the severity of the abnormality (i.e., grade) and the amount of tissue affected by the abnormality (i.e. stage). Thus each of the 3 levels had a minimum score of 0 and maximum possible score of 24, and a possible total grade or stage score of 72 for a maximum combined score of 144. Combined total score ratio (TSR) =(proximal TSR + mid TSR + distal TSR)/N, where N is the number of non missing sections for TSR. A negative change from baseline indicates that epithelial inflammation decreased.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 12 and Week 36
Population: as for outcome 13
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
score on scale
  Combined Grade TSR: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Combined Grade TSR: Week 12 | -0.1 (0.04) | -0.2 (0.03) | -0.2 (0.02) | -0.3 (0.02)
  Combined Grade TSR: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Combined Grade TSR: Week 36 | -0.2 (0.03) | -0.2 (0.04) | -0.1 (0.02) | -0.2 (0.03)
  Combined Stage TSR: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Combined Stage TSR: Week 12 | -0.1 (0.04) | -0.2 (0.03) | -0.2 (0.02) | -0.2 (0.02)
  Combined Stage TSR: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Combined Stage TSR: Week 36 | -0.2 (0.03) | -0.2 (0.03) | -0.1 (0.02) | -0.2 (0.02)

16. Secondary Outcome: Change From Current Study (SHP621-302 [NCT02736409]) Baseline in the Histopathologic Epithelial Features Combined Total Score (Grade and Stage) at Week 12 and Week 36
Description: as for outcome 15
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 12 and Week 36
Population: as for outcome 14
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
score on scale
  Combined Grade TSR: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Combined Grade TSR: Week 12 | 0.2 (0.05) | 0.0 (0.02) | 0.0 (0.01) | -0.2 (0.02)
  Combined Grade TSR: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Combined Grade TSR: Week 36 | 0.1 (0.03) | 0.1 (0.03) | 0.0 (0.02) | -0.2 (0.03)
  Combined Stage TSR: Week 12: number analyzed (Participants) | 20 | 24 | 91 | 57
  Combined Stage TSR: Week 12 | 0.2 (0.05) | 0.0 (0.02) | 0.0 (0.01) | -0.2 (0.02)
  Combined Stage TSR: Week 36: number analyzed (Participants) | 19 | 22 | 80 | 52
  Combined Stage TSR: Week 36 | 0.1 (0.03) | 0.1 (0.03) | 0.0 (0.02) | -0.2 (0.03)

17. Secondary Outcome: Proportion of Participants Who Had Greater Than or Equal to (>or=) 50 Percent (%) Reduction in DSQ Combined Score From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 12 and Week 36
Description: Dysphagia symptom response from the baseline of SHP621-301, was defined as >or=50% reduction in DSQ combined score (questions [Q] 2+3) from baseline of the induction study at Week 12 and 36 of current study. DSQ contained 4Q, all participants used diary, and responded to Q1(did you eat solid food) and Q2(didfood passslowly or get stuck). If participant's answer to Q2 was 'No', then diary ended for that day. If a participant answered 'Yes', he/she advanced to Q3(did you have to do anything to make food go down or get relief) and 4(extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0-84, with higher values representing a worse outcome. Anegative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.52 | 0.80 | 0.41 | 0.52
  Week 36 | 0.74 | 0.76 | 0.41 | 0.57

18. Secondary Outcome: Proportion of Participants Who Had Greater Than or Equal to (>or=) 50 Percent (%) Reduction in DSQ Combined Score From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 12 and Week 36
Description: Dysphagia symptom response from the baseline of SHP621-302, was defined as >or=50% reduction in DSQ combined score (questions 2+3) from baseline of the induction study at Week 36 of current study. DSQ contained 4Q, all participants used diary, and responded to Q1 (did you eat solid food) and Q2 (did food pass slowly or get stuck). If participant's answer to Q2 was 'No', then diary ended for that day. If a participant answered 'Yes', he/she advanced to Q3 (did you have to do anything to make food go down or get relief) and 4(extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0-84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.13 | 0.36 | 0.19 | 0.37
  Week 36 | 0.30 | 0.36 | 0.19 | 0.38

19. Secondary Outcome: Change in the DSQ Combined Score (Questions 2+3) From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: DSQ contain 4 questions (Q), all participants used a diary, responded to Q1 (did you eat solid food), Q2 (did food pass slowly or get stuck). If participant's answer to Q2 was 'No', then diary ended for that day. If participant answered 'Yes', he/she advanced to Q3 (did you have to do anything to make food go down or get relief), Q4 (extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ] × 14)/Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q3. Scale range for DSQ combined score was 0-84. Higher values representing a worse outcome. A Negative change from baseline indicates symptoms decreased.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 51
score on scale | -19.40 (3.627) | -23.28 (2.477) | -15.35 (1.673) | -17.33 (2.269)

20. Secondary Outcome: Change in the DSQ Combined Score (Questions 2+3) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: DSQ contain 4 questions, all participants used a diary, responded to Q1 (did you eat solid food), Q2 (did food pass slowly or get stuck). If participant's answer to Q2 was 'No', then diary ended for that day. If participant answered 'Yes', he/she advanced to Q3 (did you have to do anything to make food go down or get relief), Q4 (extent to which participant experienced pain while swallowing). DSQ combined score= ([sum of points from Q2+3 in daily DSQ] × 14)/Number of diaries reported with non-missing data. Scale range was 0-2 for Q2 and 0-4 for Q3. Scale range for DSQ combined score was 0-84. Higher values representing a worse outcome. A Negative change from baseline indicates symptoms decreased. Change in DSQ combined score (Questions 2+3) from baseline of current study at Week 36 was reported.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 46
score on scale | -4.00 (1.928) | -3.84 (1.682) | -4.39 (1.356) | -10.24 (2.183)

21. Secondary Outcome: Percent Change in the DSQ Combined Score (Questions 2+3) From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: Percent change in DSQ combined score from Induction Study (SHP621-301 [NCT02605837]) baseline to current study (SHP621-302 [NCT02736409]) final treatment period (Week 36) was reported.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 51
percent change | -79.56 (7.370) | -79.77 (6.195) | -55.82 (5.048) | -61.44 (8.653)

22. Secondary Outcome: Percent Change in the DSQ Combined Score (Questions 2+3) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: Percent change in DSQ combined score from baseline to final treatment period (Week 36) of current study was reported.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: FAS consisted of all randomized participants who received at least 1 dose of investigational product in the SHP621-302 (NCT02736409) study. Here the number of participants analyzed signifies participants whose baseline DSQ combined score was not zero. Percent change cannot be calculated if baseline DSQ combined score is zero.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 14 | 16 | 56 | 39
percent change | -47.00 (15.371) | -40.78 (19.216) | -10.18 (16.050) | -39.04 (21.413)

23. Secondary Outcome: Proportion of Participants Who Had Overall Binary Response I From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 12 and Week 36 of Current Study
Description: Overall binary response I was defined as if participant had peak eosinophil count of <=6/HPF across all esophagus levels and achieved a minimum of 30% reduction in DSQ combined score from baseline of the induction study (SHP621-301 [NCT02605837]) at Week 12 and Week 36. DSQ combined score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2 and 0 - 4 for question 3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0 - 84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: FAS included all randomized participants who received at least one dose of a SHP621-302 (NCT02736409) investigational product.
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.04 | 0.64 | 0.15 | 0.42
  Week 36 | 0.26 | 0.48 | 0.13 | 0.28

24. Secondary Outcome: Proportion of Participants Who Had Overall Binary Response I From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 12 and Week 36
Description: Overall binary response I was defined as if participant had peak eosinophil count of <=6/HPF across all esophagus levels and achieved a minimum of 30% reduction in DSQ combined score from baseline at Week 12 and Week 36. DSQ combined score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2 and 0 - 4 for question 3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0 - 84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.00 | 0.32 | 0.05 | 0.29
  Week 36 | 0.09 | 0.20 | 0.06 | 0.17

25. Secondary Outcome: Proportion of Participants Who Had Overall Binary Response II From Induction Study SHP621-301 (NCT02605837) Baseline at Week 12 and Week 36 of Current Study
Description: Overall binary response II was defined as if participant had peak eosinophil count of <=6/HPF across all esophagus levels and achieved a minimum of 50% reduction in DSQ combined score from baseline of the SHP621-301 study at Week 12 and Week 36. DSQ combined score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2 and 0 - 4 for question 3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0 - 84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.04 | 0.64 | 0.12 | 0.38
  Week 36 | 0.26 | 0.44 | 0.12 | 0.28

26. Secondary Outcome: Proportion of Participants Who Had Overall Binary Response II From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 12 and Week 36
Description: Overall binary response II was defined as if participant had peak eosinophil count of <=6/HPF across all esophagus levels and achieved a minimum of 30% reduction in DSQ combined score from baseline at Week 12 and Week 36. DSQ combined score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2 and 0 - 4 for question 3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0 - 84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Week 12 and Week 36
Population: as for outcome 4
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
proportion of participants
  Week 12 | 0.00 | 0.28 | 0.04 | 0.26
  Week 36 | 0.04 | 0.20 | 0.06 | 0.17

27. Secondary Outcome: Change in the DSQ + Pain Score (Questions 2+3+4) From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ + pain score was calculated by summing the scores of responses to questions 2, 3, and 4 by using following formula: DSQ + pain score= ([sum of points from questions 2+3+4 in the daily DSQ] ×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2, 0 - 4 for question 3 and 0 - 4 for question 4, with higher values representing a worse outcome. Scale range for DSQ + pain score was 0 - 140, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 51
score on scale | -25.86 (5.023) | -31.10 (4.015) | -21.25 (2.299) | -23.17 (3.221)

28. Secondary Outcome: Change in the DSQ+ Pain Score (Questions 2+3+4) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: DSQ contained 4 questions, all participants used a diary, and responded to Questions (Q) 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Q2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Q3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ + pain score was calculated by summing the scores of responses to Questions 2, 3, and 4. Question 1 was excluded from the DSQ + pain score. DSQ + pain score=(Sum of points from questions 2+3+4 in the daily DSQ)*14 Days/Number of dairies reported with non-missing data. Scale range was 0 - 2 for Q2, 0 - 4 for Q3 and 0 - 4 for Q4, with higher values representing a worse outcome. Scale range for DSQ + pain score was 0 - 140, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 46
score on scale | -5.67 (2.704) | -4.23 (2.003) | -5.59 (1.825) | -14.12 (2.944)

29. Secondary Outcome: Change in the DSQ Pain Score (Question 4) From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ pain score was calculated by summing the scores of responses to Question 4 only. DSQ pain score=(sum of points from questions 4 in the daily DSQ)*14 days/Number of diaries reported with non-missing data. Scale range was 0 - 4 for question 4, with higher values representing a worse outcome. Scale range for DSQ pain score was 0 - 56, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 51
score on scale | -6.46 (1.667) | -7.92 (2.130) | -5.90 (0.907) | -5.83 (1.356)

30. Secondary Outcome: Change in the DSQ Pain Score (Question 4) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: as for outcome 29
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: as for outcome 19
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 20 | 22 | 73 | 46
score on scale | -1.67 (1.039) | -0.39 (0.495) | -1.20 (0.634) | -3.88 (1.101)

31. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE's)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that started or deteriorated on or after the date of the first dose of double-blind IP in SHP621-302 and through the safety follow-up contact, or 31 days after the last dose of IP for participants who did not have a safety follow-up contact.
Time Frame: From start of the study drug administration up to follow up (Week 40)
Population: Safety Set consisted of all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 23 | 25 | 106 | 65
Participants | 14 | 21 | 72 | 49

32. Secondary Outcome: Change in DXA (Dual-Energy X-ray Absorptiometry) Imaging Results (Location: Lumbar Spine [L1-L4]) From Induction Study (SHP621-301 [NCT02605837]) Baseline at Week 36 of Current Study
Description: The sites for DXA measurement were the lumber spine (L1-L4 preferred) and total body less head. DXA scans for bone mineral density (BMD) and body composition measurements were done only for adolescent participants aged 11-17 years based on the age group in the SHP621-301 study and were completed throughout the SHP621-302 study even if participants turned 18 years. Baseline of SHP621-301 is determined at Week 0 in the SHP621-301 study. Here in this outcome measure DXA measurement of L1-L4 were reported. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: Safety set consisted of all participants who received at least 1 dose of investigational product. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 0 | 2 | 12 | 8
Z score |  | -0.185 (0.2475) | 0.020 (0.3637) | 0.100 (0.4247)

33. Secondary Outcome: Change in DXA Imaging Results (Location: Lumbar Spine [L1-L4]) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: The sites for DXA measurement were the lumber spine (L1-L4 preferred) and total body less head. DXA scans for bone mineral density (BMD) and body composition measurements were done only for adolescent participants aged 11-17 years based on the age group in the SHP621-301 study and were completed throughout the SHP621-302 study even if participants turned 18 years. Here in this outcome measure DXA measurement of L1-L4 were reported. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 0 | 2 | 12 | 8
Z score |  | -0.240 (0.7495) | 0.062 (0.4839) | 0.071 (0.4783)

34. Secondary Outcome: Change in DXA Imaging Results (Location: Whole Body) From Baseline of Induction Study (SHP621-301 [NCT02605837]) at Week 36 of Current Study
Description: The sites for DXA measurement were the lumber spine (L1-L4 preferred) and total body less head. DXA scans for bone mineral density (BMD) and body composition measurements were done only for adolescent participants aged 11-17 years based on the age group in the SHP621-301 study and were completed throughout the SHP621-302 study even if participants turned 18 years. Baseline of SHP621-301 is determined at Week 0 in the SHP621-301 study. Here in this outcome measure DXA measurement of whole body (except head) were reported. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline of induction study (SHP621-301 [NCT02605837]), Week 36
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 0 | 2 | 12 | 8
Z score |  | 0.190 (0.0424) | -0.023 (0.4510) | 0.244 (0.5543)

35. Secondary Outcome: Change in DXA Imaging Results (Location: Whole Body) From Current Study (SHP621-302 [NCT02736409]) Baseline at Week 36
Description: The sites for DXA measurement were the lumber spine (L1-L4 preferred) and total body less head. DXA scans for bone mineral density (BMD) and body composition measurements were done only for adolescent participants aged 11-17 years based on the age group in the SHP621-301 study and were completed throughout the SHP621-302 study even if participants turned 18 years. Here in this outcome measure DXA measurement of whole body (except head) were reported. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline of Current Study (SHP621-302 [NCT02736409]), Week 36
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
Number analyzed (Participants) | 0 | 2 | 12 | 8
Z score |  | 0.065 (0.0636) | -0.070 (0.4060) | 0.140 (0.4173)

36. Other Pre Specified Outcome: Proportion of Participants Who Had a Histologic Response (Eosinophil Count of Greater Than or Equal to (>or=15)/High-Powered Field [HPF]) Before or at Week 12 and Before or at Week 36
Description: Eosinophil histology relapse was defined as an eosinophil count of >or=15 eos/HPF from at least 2 of 3 levels of the esophagus.
Time Frame: Week 12 and Week 36
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group
Number analyzed (Participants) | 23 | 25
proportion of participants
  Histologic Relapse before or at Week 12 | 0.65 | 0.12
  Histologic Relapse before or at Week 36 | 0.78 | 0.36

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to follow up (Week 40)
Arm/Group | Full Responder BOS-PBO Group | Full Responder BOS-BOS Group | Non-Responder BOS-BOS Group | PBO-BOS Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/106 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/25 | 6/106 | 5/65
Other Adverse Events (participants affected / at risk) | 9/23 | 10/25 | 26/106 | 18/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Responder BOS-PBO Group (N=23) | Full Responder BOS-BOS Group (N=25) | Non-Responder BOS-BOS Group (N=106) | PBO-BOS Group (N=65)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Responder BOS-PBO Group (N=23) | Full Responder BOS-BOS Group (N=25) | Non-Responder BOS-BOS Group (N=106) | PBO-BOS Group (N=65)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 9 (11) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (18) | 1 (1)
Fatigue (General disorders) | 2 (4) | 2 (3) | 2 (2) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 6 (7) | 3 (3)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 9 (9) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Blood cortisol decreased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 4 (5)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02736409/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT02736409/SAP_001.pdf